CLINICAL TRIAL: NCT06669624
Title: Leveraging Scientific Advances to Strengthen the Implementation, Evaluation, and Impacts of Intervention Programs for Children Experiencing Early Life Adversity
Brief Title: Resilience Through Interventions for Successful Early Outcomes
Acronym: RISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of California, San Francisco (Other); The Duke Endowment (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 24-0889
Record Dates: First submitted 2024-10-28; First posted 2024-11-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Parenting Intervention; Stress; Caregiver Child Relationship; Child Behavior Problem; Mental Health
Keywords: Attachment and Biobehavioral CatchUp; Parenting Intervention; RISE study; Child behavior; Biomarkers
MeSH Terms: conditions — Psychological Well-Being; Child Behavior | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: RCT with a waitlist control group
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABC Program - no wait (Experimental): Participants immediately receive the home-based ABC, which targets parenting sensitivity and nurturance.
  Interventions: Behavioral: Attachment and Biobehavioral Catch-up (ABC)
- Waitlist-Control (ABC after delay) (Other): Participants will be placed on a four-month waitlist and then receive ABC in the same manner as the Experimental Group
  Interventions: Behavioral: Attachment and Biobehavioral Catch-up (ABC); Other: Waitlist with 4-month delay, then ABC

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch-up (ABC) — 10-session home visiting intervention designed to increase parental sensitivity and nurturance and decrease parental frightening behavior.
Other: Waitlist with 4-month delay, then ABC — A 4-month waitlist period, after which they will also receive the home-based ABC program (same as Intervention group).
  Arms: Waitlist-Control (ABC after delay)

SUMMARY:
Purpose: The purpose of this research is to determine the effects of Attachment and Biobehavioral Catch-up (ABC), an evidence-based parenting program, on stress biomarkers in children.

Participants: The study will involve approximately 150 caregiver-child dyads, with children aged between 24 and 42 months. Participants will include primary caregivers fluent in English or Spanish, along with their children who have experienced social risk factors for adversity.

Procedures (Methods): Participants will be randomly assigned to either receive the ABC parenting program (10 sessions) immediately or be placed on a wait-list, receiving the program after about 4 months. The study procedures include caregivers completing online surveys, engaging in play-based observational tasks with their children, and collecting non-invasive biological samples (saliva, cheek swab, hair) from the children and saliva samples from the caregivers at 2-3 time-points.

ELIGIBILITY:
Parent/Caregiver Inclusion Criteria :

* Aged 18 or older
* Speaks English or Spanish
* Is the parent or legal guardian with legal custody of a child aged between 24 months and 42 months
* Is a primary caregiver/parent
* Has a home-like environment in which to participate in the intervention

Child Inclusion Criteria:

* Aged between 24 months and 42 months at enrollment
* Lives with the parent/caregiver at least 50% of the time
* Has experienced social risk factors, including low income, community or family violence, previous trauma/adversity exposure, prolonged separation from caregiver, significant difficulties in relationship with caregiver Child Exclusion Criteria
* Has a diagnosed genetic or congenital disorders, including but not limited to Down syndrome, cerebral palsy, seizure disorders, endocrine disorders (or is using steroid medications, including human growth hormone), or was born with birth defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Child inflammation | Pre-intervention baseline
  Pediatric saliva samples will be assayed for cytokine concentrations.
Child inflammation | 13-20 weeks after baseline
  Pediatric saliva samples will be assayed for cytokine concentrations.
Child epigenetic age acceleration | Pre-intervention baseline
  Pediatric buccal swabs will be assayed for DNAm, which will be used to calculate child epigenetic age
Child epigenetic age acceleration | 13-20 weeks after baseline
  Pediatric buccal swabs will be assayed for DNAm, which will be used to calculate child epigenetic age
Child telomere length | Pre-intervention baseline
  DNA will be extracted from child buccal swabs to calculated T/S ratios.
Child telomere length | 13-20 weeks after baseline
  DNA will be extracted from child buccal swabs to calculated T/S ratios.
Child hair cortisol | Pre-intervention baseline
  Several strands of hair will be collected and assayed to obtain hair cortisol concentration
Child hair cortisol | 13-20 weeks after baseline
  Several strands of hair will be collected and assayed to obtain hair cortisol concentration
Child stress hormones | Pre-intervention baseline
  Child hair and saliva samples for cortisol, cortisone, DHEA, progesterone, and endocannabinoid levels to examine both cumulative and dynamic stress hormone responses.
Child stress hormones | 13-20 weeks after baseline
  Child hair and saliva samples for cortisol, cortisone, DHEA, progesterone, and endocannabinoid levels to examine both cumulative and dynamic stress hormone responses.
Parenting | Pre-intervention baseline
  Behavioral coding of parenting will be conducted using video recordings of tasks from the Early Regulation in Context Assessment.
Parenting | 13-20 weeks after baseline
  Behavioral coding of parenting will be conducted using video recordings of tasks from the Early Regulation in Context Assessment.
Child wellbeing | Pre-intervention baseline
  Caregiver reports of their child's quality of life will be obtained using the Pediatric Quality of Life (PedsQL) Inventory. Scores range from 0 to 100, with higher scores indicating better functioning.
Child wellbeing | 13-20 weeks after baseline
  Caregiver reports of their child's quality of life will be obtained using the Pediatric Quality of Life (PedsQL) Inventory. Scores range from 0 to 100, with higher scores indicating better functioning.
Child executive functioning | Pre-intervention baseline
  Child executive functioning will be assessed using the Minnesota Executive Function Scale™ The MEFS has been nationally normed based on the child's age and standardized scores are automatically generated using an algorithm that combines accuracy and response time (M = 100, SD = 15). Scores range from 60-140, with higher scores indicating better performance.
Child executive functioning | 13-20 weeks after baseline
  Child executive functioning will be assessed using the Minnesota Executive Function Scale™ The MEFS has been nationally normed based on the child's age and standardized scores are automatically generated using an algorithm that combines accuracy and response time (M = 100, SD = 15). Scores range from 60-140, with higher scores indicating better performance.
Child mental health | Pre-intervention baseline
  Child mental health will be assessed using caregiver reports through the Child Behavior Checklist preschool-aged form (1.5-5). We will use the total, internalizing, and externalizing subscales, with scores ranging from 0-200, 0-72, and 0-48, respectively. Higher scores represent worse functioning.
Child mental health | 13-20 weeks after baseline
  Child mental health will be assessed using caregiver reports through the Child Behavior Checklist preschool-aged form (1.5-5). We will use the total, internalizing, and externalizing subscales, with scores ranging from 0-200, 0-72, and 0-48, respectively. Higher scores represent worse functioning.
Caregiver anxiety | Pre-intervention baseline
  Caregiver anxiety symptoms will be assessed using the Generalized Anxiety Disorder 7-item (GAD-7) scale. The total score ranges from 0-21, with higher scores indicating more severe anxiety.
Caregiver anxiety | 13-20 weeks after baseline
  Caregiver anxiety symptoms will be assessed using the Generalized Anxiety Disorder 7-item (GAD-7) scale. The total score ranges from 0-21, with higher scores indicating more severe anxiety.
Caregiver depression | Pre-intervention baseline
  Caregiver depression symptoms will be assessed using the Patient Health Questionnaire-9 item form. Scores range from 0 to 27, with higher scores representing worse functioning.
Caregiver depression | 13-20 weeks after baseline
  Caregiver depression symptoms will be assessed using the Patient Health Questionnaire-9 item form. Scores range from 0 to 27, with higher scores representing worse functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Roubinov, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results, as well as derived data supporting the results.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: beginning 9 to 36 months following publication
Access Criteria: Investigators who propose to use the data and have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execute a data use/sharing agreement with UNC.

REFERENCES:
- [Background] McEwen LM, O'Donnell KJ, McGill MG, Edgar RD, Jones MJ, MacIsaac JL, Lin DTS, Ramadori K, Morin A, Gladish N, Garg E, Unternaehrer E, Pokhvisneva I, Karnani N, Kee MZL, Klengel T, Adler NE, Barr RG, Letourneau N, Giesbrecht GF, Reynolds JN, Czamara D, Armstrong JM, Essex MJ, de Weerth C, Beijers R, Tollenaar MS, Bradley B, Jovanovic T, Ressler KJ, Steiner M, Entringer S, Wadhwa PD, Buss C, Bush NR, Binder EB, Boyce WT, Meaney MJ, Horvath S, Kobor MS. The PedBE clock accurately estimates DNA methylation age in pediatric buccal cells. Proc Natl Acad Sci U S A. 2020 Sep 22;117(38):23329-23335. doi: 10.1073/pnas.1820843116. Epub 2019 Oct 14. PMID 31611402
- [Background] Sullivan ADW, Roubinov D, Norona-Zhou AN, Bush NR. Do dyadic interventions impact biomarkers of child health? A state-of-the-science narrative review. Psychoneuroendocrinology. 2024 Apr;162:106949. doi: 10.1016/j.psyneuen.2023.106949. Epub 2023 Dec 27. PMID 38295654
- [Background] Shonkoff JP, Boyce WT, Bush NR, Gunnar MR, Hensch TK, Levitt P, Meaney MJ, Nelson CA, Slopen N, Williams DR, Silveira PP. Translating the Biology of Adversity and Resilience Into New Measures for Pediatric Practice. Pediatrics. 2022 Jun 1;149(6):e2021054493. doi: 10.1542/peds.2021-054493. PMID 35535547
- [Background] Dozier M, Peloso E, Lewis E, Laurenceau JP, Levine S. Effects of an attachment-based intervention on the cortisol production of infants and toddlers in foster care. Dev Psychopathol. 2008 Summer;20(3):845-59. doi: 10.1017/S0954579408000400. PMID 18606034
- [Background] Dozier, M., Bernard, K., Roben, C. K., Steele, H., & Steele, M. (2017). Attachment and biobehavioral catch-up. Handbook of attachment-based interventions, 27-49.
- [Background] de Mendonca Filho EJ, Pokhvisneva I, Maalouf CM, Parent C, Mliner SB, Slopen N, Williams DR, Bush NR, Boyce WT, Levitt P, Nelson CA, Gunnar MR, Meaney MJ, Shonkoff JP, Silveira PP; JPB Research Network on Toxic Stress. Linking specific biological signatures to different childhood adversities: findings from the HERO project. Pediatr Res. 2023 Aug;94(2):564-574. doi: 10.1038/s41390-022-02415-y. Epub 2023 Jan 17. PMID 36650307